CLINICAL TRIAL: NCT04193514
Title: Brief Acceptance-based Therapy for Pregnant Women With High-risk Pregnancy
Brief Title: ACT for High-risk Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southern Methodist University (Other)
Responsible Party: Principal Investigator, Heather McClary, Director of Research Compliance, Southern Methodist University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H19-102-TUNN
Record Dates: First submitted 2019-12-06; First posted 2019-12-10 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Acceptance and Commitment Therapy
MeSH Terms: interventions — Acceptance and Commitment Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acceptance and Commitment Therapy (Experimental)
  Interventions: Other: Acceptance and Commitment Therapy
- Treatment as Usual (No Intervention)

INTERVENTIONS:
Other: Acceptance and Commitment Therapy — The intervention is a 7-day self-guided acceptance-based intervention using a published Acceptance and Commitment Therapy self-help work book. This therapy is based on the theory that rigid attempts to control internal states, thoughts and feelings, and other forms of experiential avoidance contribute to symptom development and maintenance of depression, anxiety and/or stress. The therapy includes two components: (a) educating patients about the exacerbation of stress and negative affect through rigid attempts at experiential avoidance, and (b) introducing acceptance and the willingness to experience pregnancy-related sensations and cognitions as an alternative to experiential control, through the practice of intentional and non-judgmental paying attention to one's thoughts, feelings, images and bodily sensations (including aversive symptoms) and learning to see thoughts as an ongoing process distinct from self rather than merely an event with literal meaning.
  Arms: Acceptance and Commitment Therapy

SUMMARY:
This study is designed to reduce the psychological distress of women with high-risk pregnancy. Women who express interest and are eligible will have the opportunity to participate in a 7-day acceptance therapy. This therapy is based on the theory that attempts to control internal states, thoughts and feelings can contribute to symptoms of depression, anxiety and/or stress. This study aims to educate women about how the willingness to experience uncomfortable pregnancy-related sensations and thoughts, rather than fighting them, can provide relief. The therapy is completed virtually, with the first therapy session done over video call with the therapist. Following, participants complete the remaining six days of therapy on their own using a work book. All women participating in the study will be asked to complete a series of self-report questionnaires before, during, and immediately following treatment, as well as twice postpartum. Participants will receive up to $60 and a work book for participation.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women with a current high-risk pregnancy.
2. Patients must be willing to engage in brief Acceptance-Commitment Therapy
3. Patients must be English-speaking.
4. Ages 18 years or older.

Exclusion Criteria:

1. Active suicidal ideation or self-harm in the past year; any previous history of suicide attempts.
2. History of bipolar disorder, psychosis, mental retardation or organic brain damage.
3. Currently using substances (alcohol, nicotine, marijuana, etc.)
4. Actively participating in psychotherapy for emotional or psychological problems from another provider

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2022-02-02 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Affect Schedule (PANAS) | 1 week
  The PANAS is a 20-item self-report measure for positive and negative affect. Answers range from 1 (very slightly/not al all) to 5 (extremely).

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS-21) | 1 week
  The DASS-21 is a 21-item self-report measure consisting of three subscales (depression, anxiety and stress). Answers range from 0 (did not apply to me at all) to 3 (applied to me very much).
Edinburgh Postnatal Depression Scale (EPDS) | 1 week
  The EPDS is a 10-item self-report measure of maternal depression. Scores range from 0 to 3, with a maximum score of 30.

OTHER OUTCOMES:
Acceptance and Action Questionnaire (AAQ-II) | 1 week
  The AAQ-II is a 7-item self-report questionnaire designed to measure psychological flexibility. Scores on this measure range from 1 (never true) to 7 (always true).

CONTACTS AND LOCATIONS:
Locations (1):
- Southern Methodist University, Dallas, Texas, United States